CLINICAL TRIAL: NCT00554723
Title: A Double Blind, Placebo Controlled, Randomized, Multicenter Study to Investigate CHInese Medicine NeuroAid Efficacy on Stroke Recovery
Brief Title: CHInese Medicine NeuroAid Efficacy on Stroke Recovery
Acronym: CHIMES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHIMES Society (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SQSTR03 - CHIMES
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Cerebral Infarction; Stroke
Keywords: Stroke; Cerebral infarct; Recovery; Double blind; Randomized; Placebo; Traditional Chinese Medicine; Neuroaid
MeSH Terms: conditions — Cerebral Infarction; Stroke | interventions — Neuroaid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): NeuroAid
  Interventions: Drug: NeuroAid
- B (Placebo Comparator): NeuroAid matched Placebo
  Interventions: Drug: NeuroAid matched Placebo

INTERVENTIONS:
Drug: NeuroAid — 4 capsules 3 times daily, for three months
  Other Names: Danqi Piantan Jiaonang (In China)
  Arms: A
Drug: NeuroAid matched Placebo — NeuroAid matched Placebo, 4 capsules 3 times daily, for three months
  Arms: B

SUMMARY:
CHIMES is a double blind, placebo controlled, randomized, multicenter study to test the hypothesis that NeuroAid is superior to placebo in reducing neurological deficit and improving functional outcome in patients with cerebral infarction of an intermediate range of severity.

DETAILED DESCRIPTION:
Stroke is a major cause of death and disability. Previous clinical studies performed in China have shown that NeuroAiD increase stroke patients'recovery in terms of neurological disability and functional outcome{Chen et al,2009}and thus may be beneficial as part of a post-stroke rehabilitation programme.

In the CHIMES study,we seek to test the hypothesis that NeuroAiD is superior to a placebo in reducing neurological deficit and improving functional outcome in patients recruited within 72 h after the ischemic stroke with intermediate range of severity {6<_NIHSS<_14}.More details of the study protocol have recently been published {Venketasubramanian et al,2009}.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged 18 years old and above (for Singapore 21 years and above as this is the legal age of consent)
* Subject is on anti-platelet therapy
* Subject is presented a pre-stroke Modified Rankin Scale inferior or equal to 1
* Female subject is eligible to participate in the trial if she is of non-childbearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post menopausal)
* Subject or his/her legally acceptable representative is willing to provide written informed consent
* Subject is presented with cerebral infarction with compatible imaging at Computed Tomography (CT) scan or Magnetic Resonance Imaging (MRI)
* Time window is less than 72 hours after symptoms onset
* Subject with cerebral infarction with intermediate severity range: 6 ≤ NIHSS ≤ 14

Exclusion Criteria:

* Subjects deemed unstable by investigator after thrombolysis treatment
* Subject has evidence of intra-cerebral hemorrhage on brain CT scan or MRI
* Subject has a rapidly improving neurological deficit
* Subject has definite indication for full-dose or long-term anticoagulation therapy
* Subject has other significant non-ischemic brain lesion which could affect function disability
* Subject has co-existing systemic diseases: terminal cancer, renal failure (creatinine > 200 μmol/L, if known), cirrhosis, severe dementia or psychosis
* Subject has participated in another clinical trial within the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2007-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Distribution modified Rankin Scale grades for all randomized subjects | 3 months

SECONDARY OUTCOMES:
NIHSS, Barthel Index, MMSE | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie Germaine Bousser, MD, Study Director — APHP Paris; Christopher Chen, MBBS, Principal Investigator — National University of Singapore
Locations (24):
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Penang General Hospital, George Town, Pulau Pinang, Malaysia
- Philippines (10):
  - Visayas Community Medical Center, Cebu City, Cebu
  - Baguio General Hospital and Medical Center, Baguio City
  - Chong Hua Hospital, Cebu
  - Davao Medical Center, Davao City
  - Brokenshire Hospital, Davao City
  - Davao Medical School Foundation, Davao City
  - West Visayas State University Hospital, Iloilo City
  - Jose Reyes Memorial Medical Center, Manila
  - University of Santo Tomas, Manila
  - Philippine General Hospital, Manila
- Singapore (4):
  - National University Hospital, Singapore, Singapore
  - National Neuroscience Institute - Tan Tock Seng Campus, Singapore, Singapore
  - Singapore General Hospital, Singapore, Singapore
  - Changi General Hospital, Singapore, Singapore
- University of Kelaniya, Ragama, Sri Lanka
- Thailand (7):
  - Chiangmai University Hospital, Muang City, Chiangmai
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Prasat Neurological Institute, Bangkok
  - Rajvithee Hospital, Bangkok
  - Thammasart Hospital, Bangkok
  - King Mongkutla Hospital, Bangkok
  - Siriraj Hospital, Bangkok

REFERENCES:
- [Background] Young SH, Zhao Y, Koh A, Singh R, Chan BP, Chang HM, Venketasubramanian N, Chen C; CHIMES Investigators. Safety profile of MLC601 (Neuroaid) in acute ischemic stroke patients: A Singaporean substudy of the Chinese medicine neuroaid efficacy on stroke recovery study. Cerebrovasc Dis. 2010;30(1):1-6. doi: 10.1159/000313398. Epub 2010 Apr 16. PMID 20395679
- [Background] Chen C, Venketasubramanian N, Gan RN, Lambert C, Picard D, Chan BP, Chan E, Bousser MG, Xuemin S. Danqi Piantang Jiaonang (DJ), a traditional Chinese medicine, in poststroke recovery. Stroke. 2009 Mar;40(3):859-63. doi: 10.1161/STROKEAHA.108.531616. Epub 2009 Jan 22. PMID 19164787
- [Background] Gan R, Lambert C, Lianting J, Chan ES, Venketasubramanian N, Chen C, Chan BP, Samama MM, Bousser MG. Danqi Piantan Jiaonang does not modify hemostasis, hematology, and biochemistry in normal subjects and stroke patients. Cerebrovasc Dis. 2008;25(5):450-6. doi: 10.1159/000126919. Epub 2008 Apr 16. PMID 18417963
- [Background] Venketasubramanian N, Chen CL, Gan RN, Chan BP, Chang HM, Tan SB, Picard D, Navarro JC, Baroque AC 2nd, Poungvarin N, Donnan GA, Bousser MG; CHIMES Investigators. A double-blind, placebo-controlled, randomized, multicenter study to investigate CHInese Medicine Neuroaid Efficacy on Stroke recovery (CHIMES Study). Int J Stroke. 2009 Feb;4(1):54-60. doi: 10.1111/j.1747-4949.2009.00237.x. PMID 19236501
- [Derived] Chen CLH, Chai JH, Pokharkar YM, Venketasubramanian N. Cost-effectiveness of MLC601 in post-stroke functional recovery compared with placebo - the CHIMES & CHIMES-E studies. BMC Health Serv Res. 2024 Sep 27;24(1):1127. doi: 10.1186/s12913-024-11618-4. PMID 39334395
- [Derived] Lee CF, Venketasubramanian N, Wong KS, Chen CL; CHIMES Study Investigators. Comparison Between the Original and Shortened Versions of the National Institutes of Health Stroke Scale in Ischemic Stroke Patients of Intermediate Severity. Stroke. 2016 Jan;47(1):236-9. doi: 10.1161/STROKEAHA.115.011657. Epub 2015 Dec 1. PMID 26628386
- [Derived] Chen CL, Venketasubramanian N, Lee CF, Wong KS, Bousser MG; CHIMES Study Investigators. Effects of MLC601 on early vascular events in patients after stroke: the CHIMES study. Stroke. 2013 Dec;44(12):3580-3. doi: 10.1161/STROKEAHA.113.003226. Epub 2013 Oct 17. PMID 24135924
- [Derived] Chen CL, Young SH, Gan HH, Singh R, Lao AY, Baroque AC 2nd, Chang HM, Hiyadan JH, Chua CL, Advincula JM, Muengtaweepongsa S, Chan BP, de Silva HA, Towanabut S, Suwanwela NC, Poungvarin N, Chankrachang S, Wong KS, Eow GB, Navarro JC, Venketasubramanian N, Lee CF, Bousser MG; CHIMES Study Investigators. Chinese medicine neuroaid efficacy on stroke recovery: a double-blind, placebo-controlled, randomized study. Stroke. 2013 Aug;44(8):2093-100. doi: 10.1161/STROKEAHA.113.002055. Epub 2013 Jun 18. PMID 23780952